CLINICAL TRIAL: NCT02706223
Title: A Cluster Randomised Trial of Pharmacy Led HCV Therapy Versus Conventional Treatment Pathways for HCV Positive Patients Receiving Daily OST in Pharmacies in Health Boards Within NHS Scotland
Brief Title: Testing and Treating Hepatitis C in Community Pharmacies
Acronym: SuperDOT-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2014GA07
Record Dates: First submitted 2016-03-04; First posted 2016-03-11 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Practice Patterns, Nurses'

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pharmacist Led (Experimental): This arm involved subjects following pathway of care and treatment delivery delivered by community pharmacists
  Interventions: Other: Pharmacist Led
- Nurse Led (Experimental): This arm involved subjects following the conventional pathway of care and treatment delivery delivered by specialist secondary care nurses
  Interventions: Other: Nurse led

INTERVENTIONS:
Other: Pharmacist Led — Trial of administering established, licensed treatments by a novel pathway, ie Community Pharmacists, which is hypothesized to improve treatment and retention in treatment of difficult to engage subjects
  Arms: Pharmacist Led
Other: Nurse led — Trial of administering established, licensed treatments by the conventional clinical care pathway, ie Specialist nurses
  Arms: Nurse Led

SUMMARY:
Hepatitis C Virus, (HCV), infection is a major health concern in the UK with up to 0.7% of the population infected. At best, 25% of those infected will clear the infection spontaneously, though for those who develop a chronic infection, they may go onto to develop liver cirrhosis or liver cancers.

The standard of care within the NHS is that patients with a history of intravenous drug use or those currently on methadone are at high risk of having HCV infection and should be offered HCV testing. Once diagnosed they can be referred to nurse led treatment pathways. Less than 10% of the methadone users are even tested for HCV and of them fewer than 20% go onto treatment regimens that successfully clear the infection despite regular interactions with heath care staff.

Pharmacists who have daily interactions with patients receiving methadone are ideally placed to deliver anti HCV therapy as they have daily contact with this client group and are well placed to advise on the drug therapy.

The SuperDOT C study will examine the impact of pharmacy led Directly Observed Therapy (DOT) for HCV treatment in patients attending Community Pharmacies in participating Health Boards within NHS Scotland. The impact of this approach will be compared with those referred to standard care pathways on how well participants clear their HCV infection.

DETAILED DESCRIPTION:
The SuperDOT-C study will evaluate a new pathway of care for patients on OST who are already receiving OST therapy on a daily basis from a pharmacist. Newer therapies for HCV have recently become much simpler to initiate and supervise with much improved effectiveness and as described below it is now proposed to extend the role of community pharmacists into initiating HCV therapy alongside the existing OST The SuperDOT-C study will utilise this existing environment and relationship to smooth the pathway into HCV therapy with co-administration of OST alongside the anti-HCV therapy under the supervision of the pharmacist compared with the established pathway of referral to another site and treatment with a nurse led ant-HCV treatment program. This new pathway may have positive effects on the movement towards HCV cure at multiple levels. The planned pathway is different to current care at each point, from testing and diagnosis through adherence to cure. In the planned pathway, the patient interacts with the pharmacist on a daily basis, as compared to intermittent interaction with a secondary care team member. The result being that the patient has a shorter care pathway, with less travelling and better access to anti-HCV treatment. The daily interaction with the pharmacy provides opportunities to assess and support the patient, provide sound advice and care, with the added benefit of being able to directly observe treatment, (DOT), thus potentially improving adherence.

ELIGIBILITY:
Inclusion Criteria:

* HCV PCR positive,
* Stable OST dose for greater than 12 weeks prior to study enrolment

Exclusion Criteria:

* Evidence of current or previous decompensated liver disease,
* Currently receiving HCV eradication treatment
* HIV infection,
* HBsAg positive with detectable HBV DNA,
* Pregnancy
* Cirrhosis or high fibrosis score
* Genotype deemed unsuitable for treatment with available study drugs
* Unable or unwilling to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Rate of Sustained Viral Response at 12 weeks, (SVR12), in pharmacy pathway compared with that of the current treatment pathway 12 weeks after completion of HCV therapy | 12 week SVR, (12 weeks post completion of HCV treatment)
  Blood test result; PCR - based measurement of levels of hepatitis C virus.

SECONDARY OUTCOMES:
Cost effectiveness of the pharmacist pathway as compared with the conventional care pathway | Span of study ie 24 months
  Health economics analysis
To determine whether the Pharmacist-led pathway compared with the Conventional Pathway leads to more people on OST being tested and initiating treatment | Span of study ie 24 months
  Comparison of rate of HCV testing rates in pharmacist pathway compared with current pathway
To explore whether adherence and persistence to HCV therapy in the pharmacy setting is at least similar to that in the Conventional pathway | Span of study ie 24 months
  Comparison of compliance rates of antiviral medications between pharmacist and conventional pathway.
To compare the acceptability of the Pharmacist-led pathway versus the conventional treatment pathway for OST clients | Span of study ie 24 months
  Compare the acceptability of the pharmacist pathway as compare to conventional pathway of care
To measure re-infection rate at 1 year after end of treatment in patients with SVR | Span of study ie 24 months
  Comparison of the rate of reinfections with HCV between pharmacist and conventional pathways
To compare the number of patients who drop out of the study between the two pathways | Span of study ie 24 months
  Comparison of subject drop out rates between pharmacist and conventional pathways

CONTACTS AND LOCATIONS:
Overall Officials: John F Dillon, MD, Principal Investigator — University of Dundee
Locations (3):
- United Kingdom (3):
  - NHS Grampian, Aberdeen
  - NHS Tayside, Dundee
  - NHS Greater Glasgow and Clyde, Glasgow

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Radley A, de Bruin M, Inglis SK, Donnan PT, Hapca A, Barclay ST, Fraser A, Dillon JF. Clinical effectiveness of pharmacist-led versus conventionally delivered antiviral treatment for hepatitis C virus in patients receiving opioid substitution therapy: a pragmatic, cluster-randomised trial. Lancet Gastroenterol Hepatol. 2020 Sep;5(9):809-818. doi: 10.1016/S2468-1253(20)30120-5. Epub 2020 Jun 8. PMID 32526210
- [Derived] Hickman M, Dillon JF, Elliott L, De Angelis D, Vickerman P, Foster G, Donnan P, Eriksen A, Flowers P, Goldberg D, Hollingworth W, Ijaz S, Liddell D, Mandal S, Martin N, Beer LJZ, Drysdale K, Fraser H, Glass R, Graham L, Gunson RN, Hamilton E, Harris H, Harris M, Harris R, Heinsbroek E, Hope V, Horwood J, Inglis SK, Innes H, Lane A, Meadows J, McAuley A, Metcalfe C, Migchelsen S, Murray A, Myring G, Palmateer NE, Presanis A, Radley A, Ramsay M, Samartsidis P, Simmons R, Sinka K, Vojt G, Ward Z, Whiteley D, Yeung A, Hutchinson SJ. Evaluating the population impact of hepatitis C direct acting antiviral treatment as prevention for people who inject drugs (EPIToPe) - a natural experiment (protocol). BMJ Open. 2019 Sep 24;9(9):e029538. doi: 10.1136/bmjopen-2019-029538. PMID 31551376
- [Derived] Radley A, de Bruin M, Inglis SK, Donnan PT, Dillon JF. Clinical effectiveness of pharmacy-led versus conventionally delivered antiviral treatment for hepatitis C in patients receiving opioid substitution therapy: a study protocol for a pragmatic cluster randomised trial. BMJ Open. 2018 Dec 14;8(12):e021443. doi: 10.1136/bmjopen-2017-021443. PMID 30552244